CLINICAL TRIAL: NCT07373366
Title: Effects of Neurobiological Therapy With Asymmetric Radio-electric Conveyer (REAC) in Diffuse Axonal Injury: a Randomized Controlled Trial.
Brief Title: Assessment of Noninvasive Neuromodulation in a Group of Traumatic Brain Injured Patients and Healthy Volunteers
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Istituto Rinaldi Fontana (Unknown)
Responsible Party: Principal Investigator, Sergio Brasil, MD, MD. PhD., University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 84791824.8.0000.0068
Record Dates: First submitted 2025-09-28; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Traumatic Brain Injury
Keywords: TRAUMATIC BRAIN INJURY; DIFFUSE AXONAL INJURY; NEUROMODULATION; RADIOELECTRIC ASSIMETRIC CONVEYER
MeSH Terms: conditions — Brain Injuries, Traumatic; Diffuse Axonal Injury

STUDY DESIGN:
Intervention Model Description: Patient selection Medical record, radiology, participation consent
  Step 1 (pre-intervention) qEEG, TCD and brain4care up to 3 days before the start of REAC sessions
  Step 2 (intervention) NPO neuromodulation (single session)
  Step 3 (intervention) NPPO-GW neuromodulation (18 sessions)
  Step 4 (post-intervention) qEEG, TCD and brain4care up to 3 days after the end of REAC sessions
  Follow-up discharge, 3m and 6m - mRankin, GOSE, DASS 21
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACTIVE (Active Comparator): Subjects undergoing active therapy
  Interventions: Device: Subjects in the intervention group receive low-frequency radioelectric therapy
- SHAM (Sham Comparator): Subjects receiving sham therapy
  Interventions: Device: Sham, the device simulates a therapy session

INTERVENTIONS:
Device: Subjects in the intervention group receive low-frequency radioelectric therapy — The intervention is based on two treatment protocols, the neuro-postural optimization in single aplication and brain-waves optimization in 18 sessions. This protocol is exclusive for the present study.
  Arms: ACTIVE
Device: Sham, the device simulates a therapy session — The device simulates a therapy session
  Arms: SHAM

SUMMARY:
Background: Severe traumatic brain injury, particularly diffuse axonal injury (DAI), often leads to lasting neurological issues. Cerebral dysfunction in DAI can be evaluated by monitoring cerebral electrical activity (CEA) through EEG. The radio electric asymmetric conveyer (REAC) is a noninvasive method designed to rebalance cellular polarity via endogenous bioelectric fields and modulate CEA. This technique may alter CEA, which can be detected using quantitative EEG (qEEG).

Objective: To assess qEEG changes following DAI and brain wave alterations after a REAC protocol in this group.

Methods: In this prospective, randomized, double-blind clinical trial, DAI patients will be assigned to active or sham groups for 19 sessions of either true or sham REAC following ICU discharge. Interventions include one Neuro Postural Optimization session and 18 NPPO-BWO-G sessions (up to four per day). The main outcome is to evaluate changes in qEEG patterns through population brain electrical mapping after REAC therapies.

DETAILED DESCRIPTION:
Traumatic brain injury (TBI) is a leading cause of death and disability globally, significantly affecting the quality of life for patients and caregivers.

In the United States, traumatic brain injury is the leading cause of death for people aged 1 to 45 and a major risk factor for morbidity and mortality in politrauma cases.

Although epidemiological data in Brazil are limited, studies indicate that TBI is a significant public health issue, primarily impacting the country's young and economically active population.

Automobile accidents and falls are primary causes of traumatic brain injury, with incidence rates highest among young adults (20 to 29 years) and individuals over 80 years old.

TBI is a highly heterogeneous condition, with multiple classification systems that emphasize distinct aspects such as the underlying mechanism of injury, clinical severity, radiological characteristics, and pathophysiological processes. These classifications play an important role in standardizing data collection, identifying prognostic factors, and informing the selection of appropriate therapeutic approaches tailored to individual cases.

From a pathophysiological perspective, traumatic brain injury (TBI) causes damage through primary lesions-direct energy transfer to the brain at trauma-and secondary effects, which involve cellular and molecular changes occurring for hours to weeks post-injury.

Diffuse axonal injury (DAI) is a type of lesion in TBI that leads to significant brain dysfunction and affects roughly 40% of patients, making it a leading cause of neurological problems in survivors.

Clinically, it is defined as a coma lasting more than 6 hours after TBI, excluding cases caused by ischemic brain injury or intracranial masses.

Detecting this condition during routine exams in TBI patients can be challenging, as DAI-related abnormalities are often missed by standard CT or MRI scans and may require advanced imaging techniques to identify structural changes in the central nervous system.

From a neurological perspective, TBI can result in a wide range of cognitive, behavioral, and sensory-motor changes that may affect the patient's quality of life. Cognition encompasses the processes involved in acquiring knowledge and includes factors such as thought, language, memory, reasoning, and task execution, which are considered important for intellectual development.

Although TBI is strongly linked to cognitive dysfunction, effective treatment remains difficult. While cognitive rehabilitation therapies have shown benefits in some studies, results are inconsistent.

Drug therapies for post-TBI cognitive disorders have proven ineffective. The limited effectiveness of conventional cognitive rehabilitation in DAI patients has led to the exploration of new therapies. Neuromodulation techniques, both invasive and noninvasive, offer promising options by targeting specific brain regions to alter activity and support recovery.

Radio-electric asymmetric conveyer (REAC) technology is a noninvasive technique that was first described by Rinaldi and Fontani. REAC neurobiological modulation with specific protocols such as neuro-postural-optimization (NPO) and neuro-psycho-physical-optimization - brain wave optimization-G (NPPO-BWO-G) is a safe, established technique with proven therapeutic benefits for various neurological and psychiatric disorders.

Given the significant brain damage and multiple disabling neurological sequelae, in severe TBI patients, combined with the limited efficacy of conventional pharmacological and cognitive rehabilitation interventions, REAC may be a promising therapeutic approach for affected patients. We will conduct a randomized clinical trial to assess REAC's effects in patients with DAI.

GOALS Primary Endpoint

• To evaluate the qEEG changes in patients with subacute/chronic DAI, following REAC neuromodulation.

Secondary Endpoint

* To evaluate the qEEG changes in adults free of neurological conditions, following REAC neuromodulation.
* To evaluate cognitive and humor changes in adults free of neurological conditions, following REAC neuromodulation.

ELIGIBILITY:
Inclusion Criteria:

* DAI diagnostic and consent for participation with the next of kin for each eligible patient

Exclusion Criteria:

* Open TBI
* History of chronic neurological conditions

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Observe if there are significant changes in the electroencephalographic pattern, compared between the groups. | Six months

SECONDARY OUTCOMES:
Observe if there are significant clinical improvement determined by the modified Rankin scale between the groups. | six months
  The modified Rankin scale has scores from 0 to 5, where 5 is the worst outcome (severe disability and remaining in bed), whereas 0 is the absence of any limitation (total recovery).
Observe if there are significant clinical improvement determined by the Glasgow outcome scale between the groups. | Six months
  The extended Glasgow outcome scale (GOSE) has scores from 1 to 8, considering upper limbs and/or lower limbs disability. 1 is the worst outcome (death), whereas 8 is the total recovery of upper limbs.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital das Clínicas da FM-USP, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rinaldi S, Mura M, Castagna A, Fontani V. (2014) Long-lasting changes in brain activation induced by a single REAC technology pulse in Wi-Fi bands. Randomized double-blind fMRI qualitative study. Sci Rep 4:5668. https://doi.org/10.1038/srep05668
- [Background] Castagna A, Rinaldi S, Fontani V, Aravagli L, Mannu P, Margotti ML. (2010) Does osteoarthritis of the knee also have a psychogenic component? Psycho-emotional treatment with a radio-electric device vs. intra-articular injection of sodium hyaluronate: an open-label, naturalistic study. Acupunct Electrother Res 35:1-16. https://doi.org/10.3727/036012910803860968
- [Background] Li S, Zaninotto AL, Neville IS, Paiva WS, Nunn D, Fregni F. (2015) Clinical utility of brain stimulation modalities following traumatic brain injury: current evidence. Neuropsychiatr Dis Treat 11:1573-1586. https://doi.org/10.2147/NDT.S65816
- [Background] Zaninotto AL, Vicentini JE, Solla DJ, Silva TT, Guirado VM, Feltrin F, de Lucia MC, Teixeira MJ, Paiva WS. (2017) Visuospatial memory improvement in patients with diffuse axonal injury (DAI): a 1-year follow-up study. Acta Neuropsychiatr 29:35-42. https://doi.org/10.1017/neu.2016.29
- [Background] Rinaldi C, Landre CB, Volpe MI, Goncalves RG, Nunes LDS, Darienso D, Cruz AV, Oliveira JD, Rinaldi S, Fontani V, Barcessat AR. Improving Functional Capacity and Quality of Life in Parkinson's Disease Patients through REAC Neuromodulation Treatments for Mood and Behavioral Disorders. J Pers Med. 2023 Jun 1;13(6):937. doi: 10.3390/jpm13060937. PMID 37373926
- [Background] Goncalves de Oliveira Cruz AV, Goes Goncalves R, Nunes L, Douglas Quaresma de Oliveira J, Lima Monteiro ES, Soares Eneias I, Guilherme Lima TC, Duarte Ferreira L, Souza Neri E, da Cunha Pena JL, Celis de Cardenas AM, Cortes Volpe MI, Filgueiras de Assis Melo MV, Rinaldi A, Pinheiro Barcessat AR. (2022) Neuro Postural Optimization Neuromodulation Treatment of Radio Electric Asymmetric Conveyer Technology on Stress and Quality of Life in Institutionalized Children in a Capital City of the Brazilian Amazon. Cureus 14:e26550. https://doi.org/10.7759/cureus.26550
- [Background] Pinheiro Barcessat AR, Nolli Bittencourt M, Duarte Ferreira L, de Souza Neri E, Coelho Pereira JA, Bechelli F, Rinaldi A. (2020) REAC Cervicobrachial Neuromodulation Treatment of Depression, Anxiety, and Stress During the COVID-19 Pandemic. Psychol Res Behav Manag 13:929-937. https://doi.org/10.2147/PRBM.S275730
- [Background] Rinaldi A, Rinaldi C, Coelho Pereira JA, Lotti Margotti M, Bittencourt MN, Barcessat ARP, Fontani V, Rinaldi S. (2019) Radio electric asymmetric conveyer neuromodulation in depression, anxiety, and stress. Neuropsychiatr Dis Treat 15:469-480. https://doi.org/10.2147/NDT.S195466
- [Background] Gennarelli TA, Spielman GM, Langfitt TW, Gildenberg PL, Harrington T, Jane JA, Marshall LF, Miller JD, Pitts LH. (1982) Influence of the type of intracranial lesion on outcome from severe head injury. J Neurosurg 56:26-32. https://doi.org/10.3171/jns.1982.56.1.0026
- [Background] de Almeida CE, de Sousa Filho JL, Dourado JC, Gontijo PA, Dellaretti MA, Costa BS. (2016) Traumatic Brain Injury Epidemiology in Brazil. World Neurosurg 87:540-547. https://doi.org/10.1016/j.wneu.2015.10.020
- [Background] Hyder AA, Wunderlich CA, Puvanachandra P, Gururaj G, Kobusingye OC. The impact of traumatic brain injuries: a global perspective. NeuroRehabilitation. 2007;22(5):341-53. PMID 18162698

DOCUMENTS (1):
  • Study Protocol (2025-10-15): https://cdn.clinicaltrials.gov/large-docs/66/NCT07373366/Prot_000.pdf